CLINICAL TRIAL: NCT04748315
Title: Recovery Kinetics After Speed-Εndurance Maintenance Training (SEMT) in Elite Male Soccer Players
Brief Title: Recovery Kinetics After Speed-Εndurance Maintenance Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Ioannis G. Fatouros, Professor, University of Thessaly
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: Recovery-Maintenance-UTH
Record Dates: First submitted 2021-01-25; First posted 2021-02-10 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Muscle Damage
Keywords: muscle damage; Eccentric exercise; Speed maintenance training; Soccer; Recovery

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SEMT(1:1) (Experimental): Participants in this arm will perform an a speed endurance maintenance training consisted of work to rest ratio 1:1.
  Interventions: Other: SEMT(1:1)
- SEMPT(1:3) (Experimental): Participants in this arm will perform an a speed endurance maintenance training consisted of work to rest ratio 1:3.
  Interventions: Other: SEMT (1:3)
- Control (No Intervention): Participants in this arm will receive no intervention

INTERVENTIONS:
Other: SEMT(1:1) — Soccer trainning protocolo will be performed on an work to rest ratio 1:1 and the trainning volume will consist of 1 set and 6 repetitions per set
  Arms: SEMT(1:1)
Other: SEMT (1:3) — Soccer trainning protocolo will be performed on an work to rest ratio 1:3 and the trainning volume will consist of 1 set and 6 repetitions per set
  Arms: SEMPT(1:3)

SUMMARY:
The purpose of this study will be to inestigate the recovery kinetics on performance, neuromuscular fatigue and muscle microtaruma that will occur after two speed-endurance maintenance training protocols in elite male soccer players. Also, this study will determine the comparison between two different speed endurance maintenance protocols in neuromuscular fatigue, muscle microtrauma indicators and performance factors. The training protocols will be differentiated in training work to rest ratio. The firts training protocol trial will comprise the work to rest ratio (1:1) and the other trial will comprise the work to rest ratio 1:3.

DETAILED DESCRIPTION:
Speed endurance maintenance training is utilized in order to improve the repeated sprint and high speed running ability of soccer players during a soccer match. Also, speed endurance maintenance training includes soccer drills which stimulate high speed and powerful actions such as changes of directions, accelerations and decelerations. However these actions are associated with eccentric component and it is known that eccentric exercises induces muscle damage microtrauma. Thus, the aim of this study will be to investigate the recovery kinetics on performance, neuromuscular fatigue and muscle microtrauma that will occur after two speed-endurance maintenance training protocols in elite male soccer players. The speed endurance maintenance training (SEMT) sessions will be differentiated in training volume and specifically in the work to rest period. Specifically, a randomized three-trial, cross-over, repeated measures design will be applied. Elite male soccer players (aged 18-35 years) will participate in the present study. Also, it is considered necessary that the participants will not suffer from any musculoskeletal injuries that will limit their ability to perform the SEMT sessions. Also the participants will not be smokers and will not consume alcohol and ergogenic nutritional supplements before and during the study.

In the first phase all participants will sign an informed consent form after they will be informed about all benefits and risks of this study and they will sign a recent historical of musculoskeletal injury or illness form. Subsequently, fasting blood samples will be collected by venipuncture using a disposable needle (10-gauge) in order to estimate muscle damage concentration markers (CK), blood lactate and inflammation markers (WBC). After, delayed onset muscle soreness (DOMS) in the knee flexors (KF) and extensors (KE) of both limbs, body weight (BW), height and body composition (DXA method) will be measured in the lab. Completing the first phase, participants will be instructed by a dietitian how to record a 7 days diet recalls estimating that the energy intake during the trials will be the same. The counter movement jump (CMJ) will be measured 24 hour after (second phase) on a force platform using two force platforms at 1000 Hz, with each foot in parallel on the two platforms providing a separate yet time-synchronized measurement of the data for each leg. During the CMJ will be measured the jump height (cm), the ground reaction force (N), the peak and mean power (W/kg), the vertical stiffness (Kvert, N/m/kg) and the peak rate of force development (RFD, N/s), while at the same time will be evaluated the change in peak and mean normalized EMG during the eccentric and concentric phases of the counter movement jump, for the vastus lateralis (VL), biceps femoris (BF), gastrocnemius (GAS), and gluteus maximus (GM) muscles. Electromyography data will be collected wirelessly at 2.000 Hz using a Myon MA-320 EMG system. The peak eccentric and concentric isokinetic torque of the knee flexors and extensors, in both limbs will be evaluated on an isokinetic dynamometer at 60°/sec. Also, the isometric peak torque of the knee extensors will be evaluated at 65o in both limbs. Also the fatigue rate during maximal voluntary isometric contraction will be estimated through the percent drop of peak torque between the first and the last three seconds of a 10-secong maximal isometric contraction. Also, the speed of 10m and 30m will be measured using light cells Chronojump system. The repeated sprint ability (RSA) (5x30m) will be measure using light cells Chronojump with 25 seconds rest in-between.

The soccer agility drill with a ball will be measured using light cells Chronojump in order to evaluate the soccer technical skills, 24 hour after. Finally, Open-circuit spirometry will be utilized for assessment of maximal oxygen consumption (VO2max) using an automated online pulmonary gas exchange system via breath-by-breath analysis during a graded exercise testing on a treadmill. The ability to recover after repeated intense exercise will be evaluated through the YO-YO Intermittent Recovery test level 2 and YO-YO Intermittent Endurance test level 2. 96 hours after, the participants are going to perform one of the two speed endurance maintenance training session randomly in the field. The SEMT(1:1) session will include 1 set, 6 repetitions per set and the work to rest ratio will be 1:1. The SEMT(1:3) session will iclude 1 set, 6 repetitions per set and the work to rest ratio will be 1:3. During the sessions will be assessed the change in Heart rate using a heart rate monitor and the field activity will be recorded using a global positiong system (GPS). The blood lactate will be evaluated immediately after each session. The DOMS indicator in the knee flexors (KF) and extensors (KE) of both limbs will be evaluated immediately after, 1h, 2h, 3h, 24h, 48h, and 72 hours after each session. The isometric peak torque of the knee extensors will be evaluated at 65° in limbs, post and at 1h, 2h and 3h, hours after each session. Also the fatigue rate during maximal voluntary isometric contraction will be estimated through the percent drop of peak torque between the first and the last three seconds of a 10-secong maximal isometric contraction.

Blood samples will be collected at 24h, 48h, and 72 hours after sessions. The counter movement jump (CMJ) will be measured immediately after the session, at 1h, 2h, 3h, at 24h, 48h and 72 hours after session on a force platform using two force platforms at 1000 Hz, with each foot in parallel on the two platforms providing a separate yet time-synchronized measurement of the data for each leg. During the CMJ will be measured the jump height (cm), the ground reaction force (N), the peak and mean power (W/kg), the vertical stiffness (Kvert, N/m/kg) and the peak rate of force development (RFD, N/s), while at the same time will be evaluated the change in peak and mean normalized EMG during the eccentric and concentric phases of the counter movement jump, for the vastus lateralis (VL), biceps femoris (BF), gastrocnemius (GAS), and gluteus maximus (GM) muscles. Electromyography data will be collected wirelessly at 2.000 Hz using a Myon MA-320 EMG system. Also, the speed of 10m and 30m will be measured using light cells Chronojump system immediately after, at 24h, 48h and 72 hours after session. Finally the RSA test will be measured at 24h, 48h and 72 hours after sessions. Α 2 - week washout period will be adapted among trials. After, the participants will perform the process until they complete the trials.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 35 years
* Active soccer players who participate on a competitive soccer level at least for 4 years(≥5 sessions per week ≥1 match per week)
* Free of chronic diseases
* Free of musculoskeletal injury
* Participants should be non-smokers

Exclusion Criteria:

* Musculoskeletal injury
* Chronic disease
* Use of alcohol, caffeine and any type of ergogenic supplements or medication before (≥ 6 months) and throughout the study.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 10 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Change in white blood cell count | At baseline, at 24, 48 and 72 hours post speed endurance maintenance protocols.
  White blood cell count will be measured using an automatic blood analyzer
Change in Creatine kinase in blood | At baseline, at 24, 48 and 72 hours post speed endurance maintenance protocols.
  Creatine kinase will be measured in plasma
Change in countermovement jump height | At baseline, post, 1, 2,3, 24, 48 and 72 hours post speed endurance maintenance protocols.
  Countermovement jump height will be measured using two force platforms at 1000Hz, with each foot in parallel on the two platforms providing a seperate yet time-synchronized measurement of the jump height for each leg
Change in ground reaction force (GRF) during countermovement jump test | At baseline, at post, at 1, 2, 3, 24, 48 and 72 hours post speed endurance maintenance protocols.
  The ground reaction force will be measured using two force platforms at 1000Hz, with each foot in parallel on the two platforms providing a seperate yet time-synchronized measurement of the jump height for each leg
Change in peak power during countermovement jump test | At baseline, post 1, 2, 3, 24, 48 and 72 hours post speed endurance maintenance protocols.
  The peak power will be measured using two force platforms at 1000Hz, with each foot in parallel on the two platforms providing a seperate yet time-synchronized measurement of the jump height for each leg
Change in mean power during countermovement jump test | At baseline, post, 1, 2, 3, 24, 48 and 72 hours post speed endurance maintenance protocols.
  The mean power will be measured using two force platforms at 1000Hz, with each foot in parallel on the two platforms providing a seperate yet time-synchronized measurement of the jump height for each leg
Change in vertical stifness during countermovement jump test | At baseline, post, 1, 2, 3, 24, 48 and 72 hours post speed endurance maintenance protocols.
  The vertical stifness will be measured using two force platforms at 1000Hz, with each foot in parallel on the two platforms providing a seperate yet time-synchronized measurement of the jump height for each leg
Change in peak rate of force development during countermovement jump test | At baseline, post, 1, 2, 3, 24, 48 and 72 hours post speed endurance maintenance protocols.
  The peak rate of force development will be measured using two force platforms at 1000Hz, with each foot in parallel on the two platforms providing a seperate yet time-synchronized measurement of the jump height for each leg
Change in peak normalized EMG during the eccentric and concentric phases of the countermovement jmp test | At baseline, post, 1, 2, 3, 24, 48 and 72 hours post speed endurance maintenance protocols.
  Electromyography data will be collected wirelessly at 2000Hz using a Myon MA-320 EMG system (Myon AG, Schwarzenberg, Switzerland) for the vastus lateralis (VL), biceps femoris (BF), gastrocnemius (GAS), and gluteus maximus (GM) muscles
Change in mean normalized EMG during the eccentric and concentric phases of the countermovement jump test | At baseline, post, 1, 2, 3, 24, 48 and 72 hours post speed endurance maintenance protocols.
  Electromyography data will be collected wirelessly at 2000Hz using a Myon MA-320 EMG system (Myon AG, Schwarzenberg, Switzerland) for the vastus lateralis (VL), biceps femoris (BF), gastrocnemius (GAS), and gluteus maximus (GM) muscles
Change in delayed onset of muscle soreness | At baseline, post, at 1, 2, 3, 24, 48 and 72 hours post speed endurance maintenance protocols.
  Muscle soreness will be assessed during palpation of the muscle belly and the distal region
Change in repeated sprint ability (RSA) | At baseline, at 24, 48 and 72 hours post speed endurance maintenance protocols.
  5 x 30 m sprints will be performed with 25 seconds rest in-between
Change in sprint time of 10m | At baseline, post, 24, 48 and 72 hours post speed endurance maintenance protocols.
  Sprint time will be assessed over a 10m distance using light cells.
Change in sprint time of 30m | At baseline, post, 24, 48 and 72 hours post speed endurance maintenance protocols.
  Sprint time will be assessed over a 30m distance using light cells.
Change in field activity during the speed-endurance mainetnance protocols | For 20 minutes during the speed endurance maintenance training day
  Field activity will be continuously recorded during both speed endurance maintenance protocols using global positioning system (GPS) technology
Change in heart rate during the speed-endurance mainetnance protocols | For 20 minutes during the speed endurance maintenance training day
  Heart rate will be continuously recorded during both speed endurance maintenance protocols using heart rate monitors
Change in isometric peak torque | At baseline, post, 1, 2, 3 and 24, 48 72 hours post speed endurance maintenance protocols.
  The isometric peak torque will be assessed on an isokinetic dyanmometer
Change in fatigue index of maximal voluntary isometric contraction (MVIC) during 10 seconds | At baseline, post, 1, 2, 3 and 24, 48 72 hours post speed endurance maintenance protocols.
  Fatigue rate during MVIC will be estimated through the percent drop of peak torque between the first and the last three seconds of a 10-second maximal isometric contaction
Change in blood lactate | At baseline and immediately post speed endurance maintenance protocols.
  The blood lactate will be measured using a lactate plus system

SECONDARY OUTCOMES:
Body weight | At baseline
  Body weight will be measured on a beam balance with stadiometer
Body height | At baseline
  Body height will be measured on a beam balance with stadiometer
Maximal oxygen consumption (VO2max) | At baseline
  Maximal oxygen consumption will be measured by open circuit spirometry via breath by breath method
Body fat | At baseline
  Body fat will be measured by using Dual-emission X-ray absorptiometry
Lean body mass | At baseline
  Lean body mass will be measured by using Dual-emission X-ray absorptiometry
Dietary intake | Over a 7 -day period at baseline
  Dietary intake will be assessed using 7 -day diet recalls
Soccer Agility drill | At baseline
  The soccer agility drill will be assesed using light cells chronojump
Yo-Yo Intermittent Recovery Test Level 2 | At baseline
  The Yo-Yo Intermittent Recovery Test Level 2 is considered as a maximal aerobic endurance fitness test, involving running between markers placed 20 meters apart, at increasing speeds, until exhaustion.
Yo-Yo Intermittent endurance Test Level 2 | At baseline
  The Yo-Yo Intermittent endurance Test Level 2 evaluates an individual's aerobic endurance fitness, involving running between markers placed 20 meters apart, at increasing speeds, until exhaustion.

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis Fatouros, Prof, Study Director — University of Thessaly
Locations (1):
- University o Thessaly, School of Physical Education and Sports Science, Trikala, Greece